CLINICAL TRIAL: NCT01487538
Title: Weight Maintenance Through Physical Activity and Social Support in Rural Middle-Aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0175-09-FB; 5P20NR011404 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2011-12-07 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): The intervention will be delivered through action plans, videos, discussion boards and health behavior tracking (weight, calories in and out, pedometer steps) to facilitate health management, resourcefulness and health status.
  Interventions: Behavioral: Videos; Behavioral: Action Plans; Behavioral: Discussion Boards; Behavioral: Health behavior tracking
- Standard Advice Group (Active Comparator): Standard advice group receives newsletters and health behavior tracking (weight) to initiate, increase, or sustain physical activity for weight maintenance.
  Interventions: Behavioral: Health behavior tracking

INTERVENTIONS:
Behavioral: Videos — Provide information on physical activity, diet, calorie tracking to support weight maintenance in rural women.
  Arms: intervention group
Behavioral: Action Plans — Online action plans will be used by subjects to set and evaluate physical activity goals
  Arms: intervention group
Behavioral: Discussion Boards — forum to exchange information and experiences
  Arms: intervention group
Behavioral: Health behavior tracking — online tracking of weight for both intervention and standard advice group. In addition, the intervention group will also track their calories in and out and their pedometer steps

SUMMARY:
The purpose of this study is to compare an technology-based weight maintenance intervention using action plans, videos discussion boards and health behavior tracking (weight, calories in and out, pedometer steps) with a technology-based standard advice group to facilitate health management, resourcefulness and health status for rural middle-aged women.

DETAILED DESCRIPTION:
The purpose of this research project is to evaluate the influence of a theory-based intervention using the Health Effects of Life Transitions for Women Model to promote maintenance of initial weight loss. The intervention will be designed to promote physical activity to prevent weight regain among an underserved and vulnerable population of rural, mid-life women. The intervention delivered through action plans, videos, discussion boards and health behavior tracking (weight, calories in and out, pedometer steps) to facilitate health management, resourcefulness and health status will be compared with the standard advice group who receives newsletters and health behavior tracking (weight) to initiate, increase, or sustain physical activity for weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

Women:

* aged 40-64 years;
* reported intentional weight loss of 5-10% of initial body weight within previous 6 months;
* residing in a rural county (population < 50,000 residents) or rural community (population less than 2,500) within driving distance of a UNMC College of Nursing campus;
* ability to communicate in English (verbal and written);
* ambulatory and can walk at least one block without the use of an assistive device, such as a cane, walker, or wheelchair;
* have access to the internet and current email account; and
* answer 'no' to all questions on the Physical Activity Readiness Questionnaire (PAR-Q) or obtain clearance from their physician to become more active.

Exclusion Criteria:

* instructed by a physician not to exercise;
* presence of chest pain, shortness of breath, or feelings of light-headedness upon exertion.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

PRIMARY OUTCOMES:
weight maintenance | baseline, 3 months, 6 months
  Weight maintenance (no significant change in weight from baseline which corresponds to a weight gain of less than 2.3 kg from baseline over the course of the study)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Hultquist, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Southeast District Health Department, Auburn, Nebraska, United States